CLINICAL TRIAL: NCT04582565
Title: Does a Regime of Manual Lymphatic Drainage Reduce the Incidence of Breast Cancer-related Lymphoedema Following Axillary Node Clearance: a Randomised Controlled Trial
Brief Title: Manual Lymphatic Drainage Versus Standard Treatment for the Prevention of Breast Cancer-related Lymphoedema in Patients Who Undergo Axillary Node Clearance
Acronym: BCRL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10/H0310/51
Record Dates: First submitted 2020-09-23; First posted 2020-10-09 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer Related Lymphoedema
Keywords: Breast Cancer; Lymphoedema; Manual lymphatic drainage; Decongestive lymphatic therapy
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Control group will have standard of care, consisting of verbal and written information on lymphoedema prevention and standard access to breast care nurse.
  Interventions: Other: Standard Care
- Combination product (Experimental): Decongestive lymphatic therapy (DLT). DLT group will involve manual lymphatic drainage with a trained manual lymphatic drainage therapist.
  Interventions: Combination Product: Decongestive lymphatic therapy (DLT)

INTERVENTIONS:
Combination Product: Decongestive lymphatic therapy (DLT) — Manual lymphatic drainage
  Arms: Combination product
Other: Standard Care
  Arms: Control group

SUMMARY:
Axillary lymph nodes are the main site of metastasis in breast cancer. If positive axillary lymph nodes are present, an axillary lymph node dissection (ALND) is usually performed. This procedure improves disease-free survival but comes with the risk of lymphoedema as a result of disrupted lymphatic channels. Breast cancer-related lymphoedema (BCRL) is associated with considerable morbidity, which is why proven measures to reduce its incidence would improve patient outcomes. We aimed to investigate whether a regime of manual lymphatic drainage and exercise, supervised by a manual lymphatic drainage therapist compared to standard care would reduce the incidence of breast cancer-related lymphoedema in patients undergoing ALND.

DETAILED DESCRIPTION:
Eligible patients were those in whom a primary operable breast cancer is diagnosed and in whom surgery is planned to include ALND. Patients with recurrent carcinoma, previous axillary surgery/radiotherapy or any previous arm/axillary pathology leading to arm volume changes will be excluded. Eligible participants will be identified at the breast multidisciplinary meeting and will be informed of the study and given a written information sheet. Patients who choose to participate will be asked to fill in a written consent form. Patients allocated to the decongestive lymphatic therapy group will undergo intervention for a total period of 3 months. This will consist of 2 visits to a qualified practitioner in Dr Vodder manual lymphatic drainage therapist, one at the start of the 3-month period and again 6 weeks later. Patients in both groups will also be instructed to perform self-MLD on a daily basis and will be taught a series of exercises to be performed on a daily basis. Compression hosiery will be fitted to be worn during the exercises.

ELIGIBILITY:
Inclusion criteria:

* Patients with a new diagnosis of primary operable breast cancer
* Surgery will involve axillary lymph node clearance

Exclusion criteria:

* Patients with recurrent breast cancer
* Patients with previous axillary surgery
* Patients with previous axillary radiotheraphy
* Patients with previous arm/axillary pathology leading to arm volume changes

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Absolute difference in arm volumes | Through study duration, approximately 36 months
  The primary outcome was the absolute difference in arm volumes between the affected and the contralateral arms.

SECONDARY OUTCOMES:
Patients adherence to the protocol stated exercises for 3 months post surgery | Through study duration, approximately 36 months
  The patient's acceptability of physiotherapy exercises will be sought via questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom